CLINICAL TRIAL: NCT04325854
Title: Risk Factors for Ectopic Pregnancy: Comparison of Fresh and Warmed Transfers. Analysis of a 10 Years, a Single Center Experience.
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: xxx/2020
Record Dates: First submitted 2020-03-13; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Ectopic Pregnancy; Assisted Reproductive Technology
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ectopic pregnancy population: The data have been collected from the Humanitas Fertility Center' Department database (ART.it) from all ART procedures (both I and II level) performed between 2009 and 2018.
  Interventions: Procedure: I and II level ART procedure

INTERVENTIONS:
Procedure: I and II level ART procedure — I level: Intrauterine insemination II level: Invitro fertilization technique; Intracytoplasmic sperm injection; Embryo transfer

SUMMARY:
Ectopic pregnancy (EP) is a leading cause of maternal death during the first trimester of pregnancy. Previous studies have reported an increased incidence of EP in Assisted reproductive technologies techniques (ART) (Clayton et al., 2006), and in particular with fresh blastocyst embryo transfer compared with warmed embryo transfer (Londra et al., 2015). In consideration of the widespread use of ART techniques in gynaecology and the high morbidity and mortality associated with EP, providing further insight into the risk factors associated with EPs in ART appears of great relevance. The objective of this study is to compare the incidences of EPs in all ART procedures (both I and II level) in a single, third level ART center throughout a 10-year period. In addition, we also aim to revise recognized EP's risk factors among patients undergoing these procedure and to evaluate their impact in determining extrauterine implantation

DETAILED DESCRIPTION:
Ectopic pregnancy (EP) remain a leading cause of maternal death during the first trimester of pregnancy. Previous studies have reported an increased incidence of EP in Assisted reproductive technologies techniques (ART) (Clayton et al., 2006), and in particular with fresh blastocyst embryo transfer compared with warmed embryo transfer (Londra et al., 2015). However a metanalysis on the topic argued that the results of many studies vary significantly within years of publishing and center locations; therefore, an accurate management strategy for patients at risk of ectopic gestation after invitro fertilization and embryo transfer (IVF-ET) procedure has not been established(V. Muller et al., 2016). In addition literature on I level ART procedures appears to be lacking. In consideration of the widespread use of ART techniques in gynaecology and the high morbidity and mortality associated with EP, providing further insight into the risk factors associated with EPs in ART appears of great relevance. Indeed, revising EP risk factors may help in reducing EP incidence in ART through the stratification of women according to their characteristics and the employment of special measures.

The objective of this study is to compare the incidences of EPs in all ART procedures (both I and II level) in a single, third level ART center throughout a 10-year period. In addition, we also aim to revise recognized EP's risk factors among patients undergoing these procedure and to evaluate their impact in determining extrauterine implantation.

ELIGIBILITY:
Inclusion Criteria:

* Women with diagnosis of EP. Ectopic pregnancy diagnosis was performed with B-hcg measurement and imaging visualization of the gestational sac outside the uterus

Exclusion Criteria:

* No case was excluded

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: We evaluated data from all women performing I level ART procedures (i.e Intrauterine insemination (IUI)) and II level ART procedures (i.e Invitro Fertilization (IVF) and Intracytoplasmic sperm injection (ICSI), Embryo transfer (ET)) from 2009 to 2018.
Sampling Method: Probability Sample
Enrollment: 27377 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
EP's incidence | 10 years
  measurement of incidences of EPs in Intrauterine insemination, in vitro fertilization, intracytoplasmic injection and embryo transfer.
comparison of EP's incidence with present risk factors | 10 years
  comparinson of EP's incidences according to the presence of recognized EP's risk factors such as advanced maternal age, tubal disease, BMI, smoking and PID., previous pelvic os abdominal surgeries, previous uterine surgeries, primary or secondary infertility.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clayton HB, Schieve LA, Peterson HB, Jamieson DJ, Reynolds MA, Wright VC. Ectopic pregnancy risk with assisted reproductive technology procedures. Obstet Gynecol. 2006 Mar;107(3):595-604. doi: 10.1097/01.AOG.0000196503.78126.62. PMID 16507930
- [Background] Londra L, Moreau C, Strobino D, Garcia J, Zacur H, Zhao Y. Ectopic pregnancy after in vitro fertilization: differences between fresh and frozen-thawed cycles. Fertil Steril. 2015 Jul;104(1):110-8. doi: 10.1016/j.fertnstert.2015.04.009. Epub 2015 May 5. PMID 25956363
- [Background] Muller V, Makhmadalieva M, Kogan I, Fedorova I, Lesik E, Komarova E, Dzhemlikhanova L, Niauri D, Gzgzyan A, Ailamazyan E. Ectopic pregnancy following in vitro fertilization: meta-analysis and single-center experience during 6 years. Gynecol Endocrinol. 2016 Oct;32(sup2):69-74. doi: 10.1080/09513590.2016.1232550. PMID 27759446